CLINICAL TRIAL: NCT00784641
Title: A Product Performance Evaluation of a Novel Contact Lens for Daily Disposable Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 496
Record Dates: First submitted 2008-10-31; First posted 2008-11-04 (Estimated); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Novel Bausch & Lomb Contact Lens (Experimental): Novel Bausch & Lomb daily disposable contact lenses
  Interventions: Device: Novel Bausch & Lomb daily disposable contact lenses
- SofLens (Active Comparator): Bausch & Lomb SofLens daily disposable contact lenses
  Interventions: Device: Bausch & Lomb SofLens daily disposable contact lenses.
- Acuvue (Active Comparator): Johnson and Johnson 1-Day Acuvue Moist contact lenses
  Interventions: Device: Johnson and Johnson 1-Day Acuvue Moist contact lenses

INTERVENTIONS:
Device: Novel Bausch & Lomb daily disposable contact lenses — Lenses to be worn and replaced daily for 2 weeks.
  Arms: Novel Bausch & Lomb Contact Lens
Device: Bausch & Lomb SofLens daily disposable contact lenses. — Lenses to be worn and replaced daily for 2 weeks.
  Arms: SofLens
Device: Johnson and Johnson 1-Day Acuvue Moist contact lenses — Lenses to be worn and replaced daily for 2 weeks.
  Arms: Acuvue

SUMMARY:
Evaluation of the clinical performance of a novel Bausch & Lomb daily disposable contact lens when compared to the currently marketed Bausch & Lomb SofLens® daily disposable contact lenses and the currently marketed Johnson and Johnson 1-Day Acuvue Moist contact lenses when worn by adapted soft contact lens wearers on a daily disposable basis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with VA correctable to 0.3 logMAR (driving vision) or better in each eye.
* Subjects must have clear central corneas and be free of any anterior segment disorders.
* Subjects must be myopic and require lens correction in both eyes.

Exclusion Criteria:

* Subjects with any systemic disease affecting ocular health.
* Subjects using any systemic or topical medications that will, in the Investigator's opinion, affect ocular physiology or lens performance.
* Subjects wearing monovision, multifocal or toric contact lenses.
* Subjects with grade 2 or greater slit lamp findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bev Barna, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Dr. James Ferrari, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 567 participants enrolled (1134 eyes).
Period: Overall Study
Arm/Group | Novel Bausch & Lomb Contact Lens | SofLens | Acuvue
Started | 189 | 189 | 189
Completed | 183 | 186 | 187
Not Completed | 6 | 3 | 2

BASELINE CHARACTERISTICS:
Population: There were 561 participants who were dispensed lenses (1122 eyes).
Groups:
- Total: Total of all reporting groups
Arm/Group | Novel Bausch & Lomb Contact Lens | SofLens | Acuvue | Total
Number analyzed (Participants) | 188 | 186 | 187 | 561
Age, Continuous [Mean (Full Range); unit: years] | 32.8 [18 to 67] | 32.5 [18 to 55] | 32.5 [18 to 63] | 32.6 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 147 | 136 | 137 | 420
  Male | 41 | 50 | 50 | 141

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Favorable Responses for the Initial Lens Performance Survey
Description: The initial lens performance survey was administered at the Screening/Dispensing Visit. Scores were captured on a scale from 0 to 100, with 100 being the most favorable score. Favorable responses were defined as scores of 80 or greater.
Time Frame: At dispensing
Population: Eyes that were dispensed contact lenses are included in the analysis population.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Novel Bausch & Lomb Contact Lens | SofLens | Acuvue
Number analyzed (Participants) | 188 | 186 | 187
Number analyzed (eyes) | 376 | 372 | 374
eyes
  Lens handling upon insertion | 340 | 293 | 326
  Burning/stinging upon insertion | 363 | 333 | 339
  Comfort | 333 | 289 | 354
  Vision | 324 | 338 | 363

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Adverse events were not coded. Therefore, source vocabulary is not applicable. There were 378 eyes dispensed the test lens, 376 eyes dispensed the SofLens, and 378 eyes dispensed the Acuvue lens, assessed for adverse events.
Arm/Group | Novel Bausch & Lomb Contact Lens | SofLens | Acuvue
Serious Adverse Events (participants affected / at risk) | 0/189 | 0/188 | 0/189
Other Adverse Events (participants affected / at risk) | 0/189 | 0/188 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.